## University of Texas at El Paso (UTEP) Institutional Review Board Minor Assent Form to Participate in a Research Study

Study Title: Retention of Whole-Body Vibration Training Effects on Ambulatory

Function in Children with Cerebral Palsy

Principal Investigator: Jeffrey Eggleston, PhD

**UTEP** Department of Kinesiology

This study is about learning what happens when you participate in a whole-body vibration training after 4-weeks and then after 12-weeks.

You are being asked to decide if you want to be in this research study because

• You are between the ages of 8-12 years old, you have a clinical diagnosis of Cerebral Palsy, and you can walk without assistance.

Your parent/guardian knows about the study, but you can decide if you want to be in it or not.

Before the study begins, you will be placed into one of two groups. One group is going to stand on a platform that shakes under your feet. This is called whole-body vibration. The other group of people will just stand on the platform while a noise from the machine plays. If you are in the group that shakes your body, you may or may not feel the platform as it shakes on your feet.

I know that to be in this study I will be asked to:

- Walk around the room without assistance
- Fill out a questionnaire about my happiness
- Wear markers on my body so cameras can track my movement
- Stand very still to test my balance
- Participate in a whole-body vibration training program for 4-weeks
  - 3 times a week for about 20 min each time
- Come back into the lab for 1 to 1.5 hours 12 weeks after the training program

I know that the first and the last session from the training program will last around 1.5 to 2 hours because we will be doing some tests before and after the whole-body vibration

Can anything bad happen to me?

• I know that I may get tired from walking or standing on the vibration plate, and if I do, I can tell Maria, Rene, or Jeff, and I can take a break.

Can anything good happen to me?

- I get to wear markers on my body, which will track my movements on a computer like a video game. After the study, I will be able to see my movements on the computer.
- I get to stand on a plate that will shake really fast under my feet.

What if I have questions about this study?

• I know that I can ask questions about this study at any time. You can call Maria, Rene, or Jeff, if I have questions later. The phone number is 915-747-6010

What if I don't want to do this or I change my mind later?

• I know that I can stop being in the study at any time without anyone being mad at me. I will not get in trouble if I stop being in the study.

I know that only the people who work on this research study will know my name but no one else will be given my name.

If you want to be in this study at this time, color or circle the happy face.

If you **do not** want to be in this study at this time, color or circle the sad face.



| A copy of this paper will be given to you. | |
|---|---|
| Witness or Mediator: ———————————————————————————————————— | Date: ——— |
| I have explained the research at a level that is understandable by the child and believe that the child understands what is expected during this study. | |
| Signature of Person Obtaining Assent: | |
| | Date |